CLINICAL TRIAL: NCT01005368
Title: Molecular Markers Of Chronic Lymphocytic Leukemia
Brief Title: Study of Biomarkers in Blood and Bone Marrow Samples From Patients With Previously Untreated Chronic Lymphocytic Leukemia
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-20203; CALGB-20203; CDR0000398201 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Leukemia
Keywords: chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — In Situ Hybridization, Fluorescence; Base Sequence; Polymerase Chain Reaction; Blotting, Western; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood and bone marrow samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Blood and bone marrow is collected at baseline, 3 months after completion of induction therapy, 2 months after completion of consolidation therapy, 1 year after completion of study treatment, and at disease relapse. Samples are analyzed by FISH for interphase cytogenetics, PCR for IgV_H mutational status, flow cytometry for surface expression of CD38 cells, western blot to assess Mcl-1, Bcl-2, BAK-1, ATM, ZAP-70, and Bar expression, and sequencing for p53 and ATM function.
  Interventions: Genetic: fluorescence in situ hybridization; Genetic: mutation analysis; Genetic: nucleic acid sequencing; Genetic: polymerase chain reaction; Genetic: western blotting; Other: flow cytometry; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: fluorescence in situ hybridization
Genetic: mutation analysis
Genetic: nucleic acid sequencing
Genetic: polymerase chain reaction
Genetic: western blotting
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer.

PURPOSE: This research study is looking at biomarkers in blood and bone marrow samples from patients with previously untreated chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the relevance of common and uncommon interphase cytogenetic abnormalities related to baseline clinical features, complete response (CR), prolonged progression-free survival (PFS), and overall survival (OS) in patients with previously untreated chronic lymphocytic leukemia.
* Determine the significance of the absence of IgV_H gene mutational status as related to the ability to predict CR, PFS, and OS in these patients.
* Correlate IgV_H gene mutational status with CD38 expression, ZAP-70 expression, over-expression of Mcl-1, BAK-1, high Mcl-1:Bax ratio, p53 mutations or dysfunction, high-risk karyotype abnormalities, and other molecular features associated with poor outcome in these patients.
* Determine the prognostic significance of over-expression of Mcl-1, BAK-1, high Mcl-1:Bax ratio, p53 mutations or dysfunction, ATM mutation, ATM expression, and other factors that disrupt apoptosis with respect to CR, prolonged PFS, and OS.
* Determine if clonal evolution occurs in these biological markers at partial response or disease relapse.

OUTLINE: This is a multicenter study.

Blood and bone marrow is collected at baseline, 3 months after completion of induction therapy, 2 months after completion of consolidation therapy, 1 year after completion of study treatment, and at disease relapse. Samples are analyzed by FISH for interphase cytogenetics, PCR for IgV_H mutational status, flow cytometry for surface expression of CD38 cells, western blot to assess Mcl-1, Bcl-2, BAK-1, ATM, ZAP-70, and Bar expression, and sequencing for p53 and ATM function.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia

  * Previously untreated disease
* Registered to receive treatment on a Cancer and Leukemia Group B protocol

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with chronic lymphocytic leukemia and were previously untreated. The patients must have also previously enrolled on a Cancer and Leukemia Group B protocol.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-10 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
complete response | Up to 10 years
prolonged progression-free survival | Up to 10 years
overall survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: John C. Byrd, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (35):
- United States (35):
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - National Naval Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - McLeod Regional Medical Center, Florence, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont